CLINICAL TRIAL: NCT05583565
Title: Effect of the Sensory Integration Approach on Balance and Motor Coordination in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Mohamed Reffat, lecturer at physical therapy faculty, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sensory integration
Record Dates: First submitted 2022-08-30; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Down Syndrome
Keywords: trisomy 21, Neurodevelopmental disorder
MeSH Terms: conditions — Down Syndrome; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): receiving sensory integration approach
  Interventions: Other: sensory integration approach
- control group (Active Comparator): receiving conventional physical therapy
  Interventions: Other: traditional physical therapy program

INTERVENTIONS:
Other: sensory integration approach — Sensory integration refers to how the nervous system receives messages from multimodal sensory information systems to maintain balance, posture, and balance by monitoring head movement and stabilizing the eyes about the environment
  Arms: study group
Other: traditional physical therapy program — conventional physiotherapy training programs such as the following: 1)Hand function training by locating the Grading of the hand and training this level until it is well developed to transfer to the next level according to 8 parameters (partner's height-shape-weight-texture -reaction time-speed-accuracy-number of trials).
  2) equilibrium training by promoting posture reaction. 3)ADL activity training (nutrition training-dressing training-toilet training). 4) Functional skill training through walking (walking on sand, weight on legs, and Climbing stairs ).
  Arms: control group

SUMMARY:
Down syndrome can be characterized by global mental and physical dysfunction or isolated gait, cognition, growth, or sensory disturbances. This study was conducted to investigate the effect of the sensory integration approach on improving balance and motor coordination in children with Down syndrome.

DETAILED DESCRIPTION:
Thirty children were enrolled in this study and randomly assigned to two groups: Group A received (sensory integration therapy program and training in physical therapy) and received group B (physical therapy training program only). Motor coordination and balance were assessed before and after exercise for all children using Bruininks - Oseretsky Test of Motor Proficiency - 2nd Edition.

ELIGIBILITY:
Inclusion Criteria:

* children with Down syndrome
* the ages of five and ten years who can walk
* their IQ is more than 75%

Exclusion Criteria:

* they had a serious neurological disorder (epilepsy), orthopedic problems, upper or lower limb surgery, vision or hearing problems, use of medications that impair behavior or attention, and suffered from advanced intellectual disability

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
balance | 6 months
  measured by using BOTS scale

SECONDARY OUTCOMES:
coordination | 6 months
  measured by using BOTS scale

CONTACTS AND LOCATIONS:
Locations (1):
- CairoU, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No